CLINICAL TRIAL: NCT06035354
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase Ib/II Clinical Study to Evaluate the Safety, Pharmacokinetics and Efficacy of AK120 in the Treatment of Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics and Efficacy of AK120 in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK120-102
Record Dates: First submitted 2023-06-02; First posted 2023-09-13 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- AK120 150 mg in phase Ib (Experimental): subcutaneous injection once a week for 4 weeks.
  Interventions: Drug: AK120
- AK120 300mg in phase Ib (Experimental): subcutaneous injection once a week for 4 weeks.
  Interventions: Drug: AK120
- Placebo Comparator: Placebo in phase Ib (Placebo Comparator): subcutaneous injection once a week for 4 weeks.
  Interventions: Drug: Placebo
- AK120 150mg in phase II (Experimental): subcutaneous injection every 2 weeks for 50 weeks.
  Interventions: Drug: AK120
- AK120 300mg in phase II (Experimental): subcutaneous injection every 2 weeks for 50 weeks.
  Interventions: Drug: AK120
- AK120 450mg in phase II (Experimental): subcutaneous injection every 2 weeks for 50 weeks.
  Interventions: Drug: AK120
- Placebo Comparator: Placebo in phase II (Placebo Comparator): subcutaneous injection every 2 weeks, then crossover to AK120 Regimen 4 and Regimen 5, subcutaneous injection at week 16, after primary endpoint evaluation.
  Interventions: Drug: Placebo
- AK120 150mg in phase II extension (Experimental): subcutaneous injection every 2 weeks for 14 weeks.
  Interventions: Drug: AK120
- AK120 300mg in phase II extension (Experimental): subcutaneous injection every 2 weeks for 14 weeks.
  Interventions: Drug: AK120
- AK120 450mg in phase II extension (Experimental): subcutaneous injection every 2 weeks for 14 weeks.
  Interventions: Drug: AK120

INTERVENTIONS:
Drug: AK120 — subcutaneous injection once a week
  Arms: AK120 150 mg in phase Ib
Drug: AK120 — subcutaneous injection once a week
  Arms: AK120 300mg in phase Ib
Drug: Placebo — subcutaneous injection once a week.
  Arms: Placebo Comparator: Placebo in phase Ib
Drug: AK120 — subcutaneous injection every 2 weeks.
  Arms: AK120 150mg in phase II
Drug: AK120 — subcutaneous injection every 2 weeks.
  Arms: AK120 300mg in phase II
Drug: AK120 — subcutaneous injection every 2 weeks.
  Arms: AK120 450mg in phase II
Drug: Placebo — subcutaneous injection every 2 weeks for 16 weeks then crossover to AK120 Regimen 4 and Regimen 5.
  Arms: Placebo Comparator: Placebo in phase II
Drug: AK120 — subcutaneous injection every 2 weeks
  Arms: AK120 150mg in phase II extension
Drug: AK120 — subcutaneous injection every 2 weeks.
  Arms: AK120 300mg in phase II extension
Drug: AK120 — subcutaneous injection every 2 weeks.
  Arms: AK120 450mg in phase II extension

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter phase Ib/II clinical study to evaluate the safety, pharmacokinetics and efficacy of AK120 in the treatment of subjects with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter phase Ib/II clinical study to evaluate the safety, pharmacokinetics and efficacy of AK120 in subjects with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with age 18 - 75 years (inclusive).
2. Atopic dermatitis (AD) diagnosed at least half an year before screening.
3. Subject with EASI score ≥16, IGA ≥ 3, BSA ≥ 10% at screening and baseline.
4. Subjects with a history of an inadequate response or medically inappropriate use of topical drug treatment within 6 months.

Exclusion Criteria:

1. Suffering from other inflammatory diseases that may affect efficacy outcomes (such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathy, mixed connective tissue disease, overlap syndrome, etc.).
2. History of exposure to active TB, and/or history or current evidence of TB infection.
3. Positive serology results at Screening for hepatitis B, hepatitis C or HIV.
4. Any history of vernal keratoconjunctivitis (VKC) or atopic keratoconjunctivitis (AKC) within 6 months before the baseline visit.
5. History of clinical parasite infection, recent or planned travel to an area with endemic parasite infection within 6 months before the Screening visit
6. Any medical or psychiatric condition, laboratory, or ECG parameter which, in the opinion of the Investigator or the Sponsor's medical monitor, would place the subject at risk, interfere with participation in the study, or interfere with the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Phase Ib | Baseline to week 12
  Incidence of treatment emergent AE . An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Phase Ib | Baseline to week 12
  T1/2 of AK120. Assessment of half-life(t1/2) of AK120.
Phase Ib | Baseline to week 12
  AUC of AK120. Assessment of Area under the curve(AUC) of AK120
Phase Ib | Baseline to week 12
  Cmax of AK120. Assessment of Peak concentration(Cmax) of AK120
Phase Ib | Baseline to week 12
  Tmax of AK120. Assessment of Time to peak(Tmax) of AK120
Phase II | at week 16
  Percentage of subjects who achieved (Eczema Area and Severity Index)EASI-75
Phase II Extension Study | Baseline to week 24
  Incidence of treatment emergent AE . An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
Phase Ib | Baseline to week 12
  Percentage of subjects with detectable anti AK120 antibodies (ADA).
Phase Ib | Baseline to week 12
  Percentage of subjects who achieved 0/1 in the Investigator's Global Assessment (IGA)(on a 6-point scale) .
  Lower score of IGA mean better outcome, higher score mean worse outcome
Phase II | Baseline to week 58
  Percentage of subjects who achieved EASI-50 (≥50% improvement from baseline) /EASI-75 (≥75% improvement from baseline) response at each visit.
  Higher score mean better outcome, lower score mean worse outcome
Phase II | Baseline to week 58
  Percentage change in EASI scores from baseline at each visit. Higher score mean better outcome, lower score mean worse outcome
Phase II Extension Study | Baseline to week 24
  Percentage of subjects who achieved EASI-50 (≥50% improvement from baseline) /EASI-75 (≥75% improvement from baseline) response at each visit.
  Higher score mean better outcome, lower score mean worse outcome
Phase II Extension Study | Baseline to week 24
  Percentage change in EASI scores from baseline at each visit. Higher score mean better outcome, lower score mean worse outcome

CONTACTS AND LOCATIONS:
Locations (39):
- China (39):
  - AkesoBio Investigative Site 2037, The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - AkesoBio Investigative Site 2036, The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - AkesoBio Investigative Site 1001, Peking University People's Hospital, Beijing, Beijing Municipality
  - AkesoBio Investigative Site 2044, Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - AkesoBio Investigative Site 2023, Xinqiao Hospital Medical University, Chongqing, Chongqing Municipality
  - AkesoBio Investigative Site 2024, Chongqing Three Gorges Medical College, Chongqing, Chongqing Municipality
  - AkesoBio Investigative Site 2040, Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - AkesoBio Investigative Site 2052, The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - AkesoBio Investigative Site 2038, The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - AkesoBio Investigative Site 2022, Dongguan People's Hospital, Dongguan, Guangdong
  - AkesoBio Investigative Site 1002, Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - AkesoBio Investigative Site 2003, Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - AkesoBio Investigative Site 2049, The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - AkesoBio Investigative Site 2004, The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - AkesoBio Investigative Site 2001, Affiliated Hospital of Chengde medical university, Chengde, Hebei
  - AkesoBio Investigative Site 2010, Nanyang First People's Hospital National Third Class A Hospital, Nanyang, Henan
  - AkesoBio Investigative Site 2051, Jingzhou Central Hospital, Jingzhou, Hubei
  - AkesoBio Investigative Site 1005, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - AkesoBio Investigative Site 2046, The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - AkesoBio Investigative Site 2008, The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - AkesoBio Investigative Site 2048, The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - AkesoBio Investigative Site 2050, Wuxi Second People's Hospital, Wuxi, Jiangsu
  - AkesoBio Investigative Site 2025, Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - AkesoBio Investigative Site 2032, The First Affiliated Hospital of Gannan Medical College, Ganzhou, Jiangxi
  - AkesoBio Investigative Site 2011, Northeast International Hospital, Shenyang, Liaoning
  - AkesoBio Investigative Site 2039, Shandong Provincial Dermatology Hospital, Jinan, Shandong
  - AkesoBio Investigative Site 2041, Qilu Hospital of Shandong University, Jinan, Shandong
  - AkesoBio Investigative Site 1003, Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - AkesoBio Investigative Site 2027, Medical School of Yanan University, Xianyang, Shanxi
  - AkesoBio Investigative Site 2029, West China Hospital，Sichuan University, Chengdu, Sichuan
  - AkesoBio Investigative Site 2034, Chengdu Second People's Hospital, Chengdu, Sichuan
  - AkesoBio Investigative Site 2013, Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - AkesoBio Investigative Site 2019, Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - AkesoBio Investigative Site 2043, First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - AkesoBio Investigative Site 1004, Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - AkesoBio Investigative Site 2006,Affiliated Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - AkesoBio Investigative Site 2007, Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - AkesoBio Investigative Site 2035, The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - AkesoBio Investigative Site 2009, The First Hospital of Jiaxing, Jiaxing, Zhejiang

IPD SHARING:
Plan to Share IPD: No